CLINICAL TRIAL: NCT00621842
Title: Open-label, Prospective Trial of Lamotrigine for Symptoms of Geriatric Bipolar Depression
Brief Title: Lamotrigine for Symptoms of Geriatric Bipolar Depression
Acronym: Geri-BD SAD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Martha Sajatovic, Professor of Psychiatry, University Hospitals Cleveland Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L0971; GSK110720; IND 78,081 (Other: FDA)
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Results first posted 2011-10-25 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Bipolar Disorder; Depression, Bipolar
Keywords: Geriatric Psychiatry; Aged; lamotrigine
MeSH Terms: conditions — Bipolar Disorder | interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open-Label Lamotrigine Treatment (Experimental)
  Interventions: Drug: Lamotrigine regular tablet formulation; Drug: Lamotrigine novel formulation

INTERVENTIONS:
Drug: Lamotrigine regular tablet formulation — Day 0 lamotrigine regular tablet formulation or lamotrigine novel formulation will be initiated at 25 mg/day and upward titrated as per package insert to targeted maximum dose of 200 mg/day. Dosing will be reduced for individuals who experience adverse effects. Dosing will be modified as per package insert for lamotrigine for individuals on anticonvulsant compounds.
  Other Names: Lamictal
Drug: Lamotrigine novel formulation — Participants will have the option of trying a novel formulation of lamotrigine tablets instead of the lamotrigine regular formulation tablets. The dosing will remain the same regardless of which type of lamotrigine tablet is used.
  Day 0 lamotrigine regular tablet formulation or lamotrigine novel formulation will be initiated at 25 mg/day and upward titrated as per package insert to targeted maximum dose of 200 mg/day. Dosing will be reduced for individuals who experience adverse effects. Dosing will be modified as per package insert for lamotrigine for individuals on anticonvulsant compounds.
  Other Names: Lamictal

SUMMARY:
This is a 12-week, open label trial of lamotrigine for older adults (age 60 and older) with type I or type II Bipolar depression. Non-demented older adults with Bipolar I or II depression, confirmed via the Structured Clinical Interview for the Diagnostic and Statistical Manual for Mental Disorders (DSM) - Patient edition (SCID-I/P) and meeting inclusion criteria for depressive symptom severity (score of 18 or greater on the Hamilton Depression Rating Scale/HAM-D-24) will receive add-on lamotrigine dosed to a target of 200 mg/day.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 Years or older
* BP Disorder-I or II: Depressive episode (DSM -IV-TR; SCID-I/P)
* HAM-D score > 18 (GRID-HAM-D 24-item version)
* Availability of an Informant is encouraged but not required for study participation

Exclusion Criteria:

* Chronic psychotic conditions, ie. schizophrenia, schizoaffective disorder, delusional disorder
* Contraindication to lamotrigine (Physician interview, medical assessment)
* Documented history of intolerance to lamotrigine
* Patients who have previously failed to respond to at least 12 weeks of treatment with lamotrigine
* Active substance dependence (SCID-I/P) or substance-related safety issues or PI concerns
* Mood Disorder Due to a General Medical Condition or Treatment (Physician interview)
* Rapid cycling (Physician interview): As defined in DSM-IV: At least 4 episodes of mood disturbance in the previous 12 months that meet criteria for a Major Depressive, Manic, Mixed or Hypomanic Episode. Episodes are distinguished either by partial or full remission for at least 2 months or by a switch to an episode of opposite polarity
* Dementia (by DSM-IV or brain degenerative diseases; Physician interview);
* Inability to communicate in English (i.e., interview cannot be conducted without an interpreter; subject largely unable to understand questions and cannot respond in English)
* Clinically significant sensory impairment (i.e., cannot see well enough to read consent or visually-presented material; cannot hear well enough to cooperate with interview; Physician interview)
* Recent history of cardiovascular, peripheral vascular events or stroke
* High risk for suicide (e.g., active SI or current intent or plan)
* Inpatient status

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2008-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha Sajatovic, MD, Principal Investigator — Case Western Reserve University School of Medicine
Locations (5):
- United States (5):
  - Weill Medical College of Cornell University, White Plains, New York
  - University Hospitals Case Medical Center/ Case Western Reserve University, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh School of Medicine, Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania
  - Baylor College of Medicine/Michael E. DeBakey VAMC, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in January 2008 and ended in December 2009. The study screened and enrolled participants at five academic institutions in the United States.
Pre-assignment Details: All subjects were required to have a score of 18 or higher on the Hamilton Rating Scale for Depression 24 to be included in the study.
Groups:
- Open-label Lamotrigine Treatment: This solitary group received open-label lamotrigine treatment for bipolar depression.
Period: Overall Study
Arm/Group | Open-label Lamotrigine Treatment
Started | 57
Completed | 38
Not Completed | 19
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 7
Not completed — Protocol Violation | 4
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Arm/Group | Open-label Lamotrigine Treatment
Number analyzed (Participants) | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 34
Region of Enrollment [Number; unit: participants]
  United States | 57

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Change in Depressive Symptoms From Baseline on the Montgomery Asberg Depression Rating Scale (MADRS)
Description: The minimum possible score is 0 and the maximum score is 60. A higher score implies a worse condition.
Time Frame: 12 weeks
Population: The number of participants for analysis was determined by number of completers plus number of dropouts where the last known observation of a dropout taking lamotrigine was carried forward. Missing data and the lack of 3 participants completing more than the baseline assessment yielded a number for analysis that was less than total enrollment.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Open-label Lamotrigine Treatment
Number analyzed (Participants) | 54
units on a scale | -15.5 [-18.0 to -12.9]
Statistical Analysis 1: Comparison: Open-label Lamotrigine Treatment; The null hypothesis is that the mean difference score between the 12 week time point or LOCF and baseline is zero; Test type: Superiority or Other; p < .01, t-test, 2 sided; df=53; Mean Difference (Final Values) = -15.5, 95% CI 2-sided [-18.0 to -12.9]

2. Secondary Outcome: Assessment of Adverse Effects With the Udvalg Fur Kliniske Undersogelser (UKU)
Description: Frequency of adverse effects was measured using the UKU. The total number of adverse effects assessed by the UKU is 49 plus one open-ended question about any adverse effects not assessed.
Time Frame: 12 weeks
Population: The number of participants was chosen from the number who received at least one dose of lamotrigine.
Measure: Number; unit: participants
Arm/Group | Open-label Lamotrigine Treatment
Number analyzed (Participants) | 57
participants
  reduced sleep duration | 14
  weight loss | 12
  increased dream activity | 12
  polyuria/polydipsia | 11
  weight gain | 9
  increased sleep | 9
  lassitude/fatigue | 8
  unsteady gait | 8

3. Secondary Outcome: Change in Depressive Symptoms From Baseline Using the Hamilton Depression Rating Scale (GRID-HAM-D)
Description: The minimum possible score is 0 and the maximum score is 78. A higher score implies a worse condition.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Open-label Lamotrigine Treatment
Number analyzed (Participants) | 54
units on a scale | -15.2 [-17.5 to -12.9]
Statistical Analysis 1: Comparison: Open-label Lamotrigine Treatment; The null hypothesis is that the mean difference score between the 12 week time point or LOCF and baseline is zero; Test type: Superiority or Other; p < .01, t-test, 2 sided; Mean Difference (Final Values) = -15.2, 95% CI 2-sided [-17.5 to -12.9]

4. Secondary Outcome: Change in Manic Symptoms From Baseline Using the Young Mania Rating Scale (YMRS)
Description: The minimum possible score is 0 and the maximum score is 60. A higher score implies a worse condition.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Open-label Lamotrigine Treatment
Number analyzed (Participants) | 49
units on a scale | -.47 [-1.82 to .88]
Statistical Analysis 1: Comparison: Open-label Lamotrigine Treatment; The null hypothesis is that the mean difference score between the 12 week time point or LOCF and baseline is zero; Test type: Superiority or Other; p = .49, t-test, 2 sided; Mean Difference (Final Values) = -.47, 95% CI 2-sided [-1.82 to .88]

5. Secondary Outcome: Change From Baseline in Overall Clinical Diagnosis Using the CGI-BP
Description: The minimum possible score is 1 and the maximum score is 7. A higher score implies a worse condition.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Open-label Lamotrigine Treatment
Number analyzed (Participants) | 53
units on a scale | -2.06 [-2.43 to -1.68]
Statistical Analysis 1: Comparison: Open-label Lamotrigine Treatment; The null hypothesis is that the mean difference between the 12 week time point or LOCF and baseline is zero; Test type: Superiority or Other; p < .01, t-test, 2 sided; Mean Difference (Final Values) = -2.06, 95% CI 2-sided [-2.43 to -1.68]

6. Secondary Outcome: Change in or Appearance of Extrapyramidal Symptoms From Baseline Using the Simpson Angus Scale (SAS)
Description: The minimum possible score is 0 and the maximum score is 4. A higher score implies a worse condition.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Open-label Lamotrigine Treatment
Number analyzed (Participants) | 48
units on a scale | -.04 [-.36 to .28]
Statistical Analysis 1: Comparison: Open-label Lamotrigine Treatment; The null hypothesis is that the mean difference between the 12 week time point or LOCF and baseline is zero; Test type: Superiority or Other; p = .80, t-test, 2 sided; Mean Difference (Final Values) = -.04, 95% CI 2-sided [-.36 to .28]

7. Secondary Outcome: Change in Body Weight From Baseline
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: lbs.
Arm/Group | Open-label Lamotrigine Treatment
Number analyzed (Participants) | 52
lbs. | .83 [-.97 to 2.62]
Statistical Analysis 1: Comparison: Open-label Lamotrigine Treatment; The null hypothesis is that the mean difference between the 12 week time point or LOCF and baseline is zero; Test type: Superiority or Other; p = .36, t-test, 2 sided; Mean Difference (Final Values) = .83, 95% CI [-.97 to 2.62]

8. Secondary Outcome: Number of Participants Who Fell at Least Once During the Study
Time Frame: 12 weeks
Population: The number of participants was chosen from the number who received at least one dose of lamotrigine.
Measure: Number; unit: participants
Arm/Group | Open-label Lamotrigine Treatment
Number analyzed (Participants) | 57
participants | 18

9. Secondary Outcome: Change in Appearance of Extrapyramidal Symptoms From Baseline Using the Abnormal Involuntary Movement Scale (AIMS)
Description: The minimum possible score is 0 and the maximum score is 4. A higher score implies a worse condition.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Open-label Lamotrigine Treatment
Number analyzed (Participants) | 48
units on a scale | -.79 [-1.67 to .09]
Statistical Analysis 1: Comparison: Open-label Lamotrigine Treatment; The null hypothesis is that the mean difference between the 12 week time point or LOCF and baseline is zero; Test type: Superiority or Other; p = .08, t-test, 2 sided; Mean Difference (Final Values) = -.79, 95% CI 2-sided [-1.67 to .09]

10. Secondary Outcome: Change in or Appearance of Extrapyramidal Symptoms From Baseline Using the Barnes Akathisia Scale (BAS)
Description: The minimum possible score is 0 and the maximum score is 5. A higher score implies a worse condition.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Open-label Lamotrigine Treatment
Number analyzed (Participants) | 47
units on a scale | -.53 [-1.03 to -.04]
Statistical Analysis 1: Comparison: Open-label Lamotrigine Treatment; The null hypothesis is that the mean difference between the 12 week time point or LOCF and baseline is zero; Test type: Superiority or Other; p = .04, t-test, 2 sided; Mean Difference (Final Values) = -.53, 95% CI [-1.03 to -.04]

11. Secondary Outcome: Number of Participants Who Had a Fall That Required Medical Attention
Time Frame: 12 weeks
Population: The number of participants was chosen from the number who received at least one dose of lamotrigine.
Measure: Number; unit: participants
Arm/Group | Open-label Lamotrigine Treatment
Number analyzed (Participants) | 57
participants | 5

12. Secondary Outcome: Number of Participants Who Had a Fall That Required Medical Attention and Was Related to Lamotrigine
Time Frame: 12 weeks
Population: The number of participants was chosen from the number who received at least one dose of lamotrigine.
Measure: Number; unit: participants
Arm/Group | Open-label Lamotrigine Treatment
Number analyzed (Participants) | 57
participants | 1

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the duration of the study (over two years) separate from any data collected using the UKU.
Arm/Group | Open-label Lamotrigine Treatment
Serious Adverse Events (participants affected / at risk) | 2/57
Other Adverse Events (participants affected / at risk) | 22/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Lamotrigine Treatment (N=57)
Hospital Admission for Increased Anxiety (Psychiatric disorders) | 1 (1)
Hospital Admission for Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Lamotrigine Treatment (N=57)
Weight gain (Metabolism and nutrition disorders) | 4 (4)
Weight Loss (Metabolism and nutrition disorders) | 4 (6)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Increased Urinary Frequency (Renal and urinary disorders) | 3 (4)
Fall (Injury, poisoning and procedural complications) | 18 (28)
Vomiting (Gastrointestinal disorders) | 4 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less